CLINICAL TRIAL: NCT04105972
Title: A Phase 3b, Randomized, Double-blind, Controlled Study Evaluating the Efficacy and Safety of VX-445/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects, Homozygous for F508del
Brief Title: A Study Evaluating the Efficacy and Safety of VX-445/Tezacaftor/Ivacaftor in Cystic Fibrosis Subjects, Homozygous for F508del
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX18-445-109; 2019-001735-31 (EudraCT Number)
Expanded Access: NCT04058210 (Approved for marketing)
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Results first posted 2021-08-18 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; tezacaftor, ivacaftor drug combination; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TEZ/IVA (Active Comparator): Following TEZ/IVA run-in period of 4 weeks, participants received TEZ 100 milligrams (mg) once daily (qd)/IVA 150 mg every 12 hours (q12h) in the treatment period for 24 weeks.
  Interventions: Drug: TEZ/IVA; Drug: IVA
- ELX/TEZ/IVA (Experimental): Following TEZ/IVA run-in period of 4 weeks, participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — FDC tablet for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
  Arms: ELX/TEZ/IVA
Drug: TEZ/IVA — Fixed-dose combination (FDC) tablet for oral administration.
  Other Names: VX-661/VX-770; tezacaftor/ivacaftor
  Arms: TEZ/IVA
Drug: IVA — Mono tablet for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
This study will evaluate the efficacy, safety, and pharmacodynamics of elexacaftor (ELX, VX-445) in triple combination (TC) with tezacaftor (TEZ) and ivacaftor (IVA) in subjects with cystic fibrosis (CF) who are homozygous for F508del.

ELIGIBILITY:
Key Inclusion Criteria:

* Homozygous for the F508del mutation (F/F)
* Forced expiratory volume in 1 second (FEV1) value ≥40% and ≤90% of predicted mean for age, sex, and height

Key Exclusion Criteria:

* Clinically significant cirrhosis with or without portal hypertension
* Lung infection with organisms associated with a more rapid decline in pulmonary status
* Solid organ or hematological transplantation

Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- Australia (6):
  - The Prince Charles Hospital, Chermside
  - Institute for Respiratory Health, Nedlands
  - Perth Children's Hospital, Nedlands
  - John Hunter Hospital & Hunter Medical Research Institute and John Hunter Children's Hospital, New Lambton
  - The Royal Children's Hospital, Parkville, VIC
  - Queensland Children's Hospital, South Brisbane
- Belgium (4):
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - UZ Antwerpen, Edegem
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Germany (8):
  - Charite Paediatric Pulmonology Department, Berlin
  - Universitaetsklinkum Koeln, CF-Studienzentrum, Cologne
  - Ruhrlandklinik Westdeutsches Lungenzentrum am Klinikum Essen, Essen
  - Universitatsklinikum Essen (AoR), Kinderklinik III, Abt. fur Pneumologie, Essen
  - Johann Wolfgang Goethe University, Frankfurt
  - Mukeviszidose-Zentrum am Universitatsklinikum Jena, Klinik fuer Kinder- und Jugendmedizin, Jena
  - Klinikum Innenstadt, University of Munich, München
  - Pneumologisches Studienzentrum Muenchen-West, München
- United Kingdom (17):
  - Belfast City Hospital, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol Royal Hospital, Bristol
  - Papworth Hospital NHS Foundation Trust, Papworth Everard, Cambridge
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter NHS Foundation Trust, Royal Devon and Exeter Hospital, Exeter
  - Clinical Research Facility, Queen Elizabeth University Hospital, Glasgow
  - St. James University Hospital, Leeds
  - Leeds General Infirmary, Leeds, West Yorkshire
  - Alder Hey Children's Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Sick Children, London
  - London and St Bartholomew's Hospital, London
  - The University Hospital of South Manchester, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, The Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Queens Medical Center, Nottingham
  - All Wales Adult Cystic Fibrosis Centre, University Hospital Llandough, Penarth
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent research/clinical-trial-data-sharing.

REFERENCES:
- [Derived] Heneghan M, Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2023 Nov 20;11(11):CD010966. doi: 10.1002/14651858.CD010966.pub4. PMID 37983082
- [Derived] Sutharsan S, McKone EF, Downey DG, Duckers J, MacGregor G, Tullis E, Van Braeckel E, Wainwright CE, Watson D, Ahluwalia N, Bruinsma BG, Harris C, Lam AP, Lou Y, Moskowitz SM, Tian S, Yuan J, Waltz D, Mall MA; VX18-445-109 study group. Efficacy and safety of elexacaftor plus tezacaftor plus ivacaftor versus tezacaftor plus ivacaftor in people with cystic fibrosis homozygous for F508del-CFTR: a 24-week, multicentre, randomised, double-blind, active-controlled, phase 3b trial. Lancet Respir Med. 2022 Mar;10(3):267-277. doi: 10.1016/S2213-2600(21)00454-9. Epub 2021 Dec 20. PMID 34942085
- [Derived] Southern KW, Murphy J, Sinha IP, Nevitt SJ. Corrector therapies (with or without potentiators) for people with cystic fibrosis with class II CFTR gene variants (most commonly F508del). Cochrane Database Syst Rev. 2020 Dec 17;12(12):CD010966. doi: 10.1002/14651858.CD010966.pub3. PMID 33331662

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 176 participants were enrolled in the study. Out of those 176 participants, 1 participant was randomized but not dosed in the treatment period. Therefore, results are presented for only 175 participants.
Pre-assignment Details: This study was conducted in cystic fibrosis (CF) participants aged 12 years or older.
Groups:
- TEZ/IVA: Following TEZ (tezacaftor)/IVA (ivacaftor) run-in period of 4 weeks, participants received TEZ 100 milligrams (mg) once daily (qd)/IVA 150 mg every 12 hours (q12h) in the treatment period for 24 weeks.
- ELX/TEZ/IVA: Following TEZ/IVA run-in period of 4 weeks, participants received ELX (elexacaftor) 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
Period: Overall Study
Arm/Group | TEZ/IVA | ELX/TEZ/IVA
Started | 88 | 87
Completed | 86 | 86
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- TEZ/IVA: Following TEZ/IVA run-in period of 4 weeks, participants received TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | TEZ/IVA | ELX/TEZ/IVA | Total
Number analyzed (Participants) | 88 | 87 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (11.0) | 27.9 (11.8) | 27.8 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 43 | 88
  Male | 43 | 44 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 83 | 85 | 168
  Unknown or Not Reported | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 0 | 2 | 2
  White | 88 | 84 | 172
  White, Asian | 0 | 1 | 1
CF Questionnaire-Revised (CFQ-R) Respiratory Domain Score [Mean (Standard Deviation); unit: units on a scale] — The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
  units on a scale | 73.1 (17.6) | 71.2 (19.6) | 72.2 (18.6)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in CF Questionnaire-Revised (CFQ-R) Respiratory Domain Score
Description: The CFQ-R is a validated participant-reported outcome measuring health-related quality of life for participants with cystic fibrosis. Respiratory domain assessed respiratory symptoms, score range: 0-100; higher scores indicating fewer symptoms and better health-related quality of life.
Time Frame: From Baseline Through Week 24
Population: Full analysis set (FAS) included all randomized participants who carried the intended CF transmembrane conductance regulator (CFTR) allele mutation and received at least 1 dose of study drug in treatment period.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | TEZ/IVA | ELX/TEZ/IVA
Number analyzed (Participants) | 88 | 87
units on a scale | 1.2 (1.5) | 17.1 (1.5)
Statistical Analysis 1: Comparison: TEZ/IVA vs ELX/TEZ/IVA; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; Least Squares (LS) Mean Difference = 15.9, 95% CI 2-sided [11.7 to 20.1]

2. Secondary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1)
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration.
Time Frame: From Baseline Through Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | TEZ/IVA | ELX/TEZ/IVA
Number analyzed (Participants) | 88 | 87
percentage points | 1.0 (0.7) | 11.2 (0.7)
Statistical Analysis 1: Comparison: TEZ/IVA vs ELX/TEZ/IVA; Test type: Superiority; p < 0.0001, Mixed-effects Model for Repeated Measure; LS Mean Difference = 10.2, 95% CI 2-sided [8.2 to 12.1]

3. Secondary Outcome: Absolute Change in Sweat Chloride (SwCl)
Description: Sweat samples were collected using an approved collection device.
Time Frame: From Baseline Through Week 24
Population: FAS.
Measure: Least Squares Mean (Standard Error); unit: millimole per liter (mmol/L)
Arm/Group | TEZ/IVA | ELX/TEZ/IVA
Number analyzed (Participants) | 88 | 87
millimole per liter (mmol/L) | -3.4 (1.2) | -46.2 (1.3)
Statistical Analysis 1: Comparison: TEZ/IVA vs ELX/TEZ/IVA; Test type: Superiority; LS Mean Difference = -42.8, 95% CI 2-sided [-46.2 to -39.3]

4. Secondary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: From Day 1 in the Treatment Period up to 28 Days After Last Dose of Study Drug or to the Completion of Study Participation Date, Whichever Occurs First (up to Week 28)
Population: Safety set included all participants who received at least 1 dose of study drug in the treatment period.
Measure: Number; unit: participants
Arm/Group | TEZ/IVA | ELX/TEZ/IVA
Number analyzed (Participants) | 88 | 87
participants
  Participants With TEAEs | 81 | 77
  Participants With SAEs | 14 | 5

ADVERSE EVENTS:
Time Frame: From Day 1 in the Treatment Period up to 28 Days After Last Dose of Study Drug or to the Completion of Study Participation Date, Whichever Occurs First (up to Week 28)
Arm/Group | TEZ/IVA | ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/88 | 0/87
Serious Adverse Events (participants affected / at risk) | 14/88 | 5/87
Other Adverse Events (participants affected / at risk) | 72/88 | 59/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEZ/IVA (N=88) | ELX/TEZ/IVA (N=87)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 1 | 0
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 9 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Type 3 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TEZ/IVA (N=88) | ELX/TEZ/IVA (N=87)
Abdominal pain (Gastrointestinal disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 8
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 32 | 10
Nasopharyngitis (Infections and infestations) | 13 | 17
Upper respiratory tract infection (Infections and infestations) | 5 | 9
Alanine aminotransferase increased (Investigations) | 1 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 5
Bacterial test positive (Investigations) | 5 | 1
Headache (Nervous system disorders) | 18 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 11
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 16 | 10
Rash (Skin and subcutaneous tissue disorders) | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04105972/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-02): https://cdn.clinicaltrials.gov/large-docs/72/NCT04105972/SAP_001.pdf